CLINICAL TRIAL: NCT01337544
Title: Haploidentical Stem Cell Transplantation and IL-15 NK Cell Infusion for Paediatric Refractory Solid Tumours
Acronym: NK
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The parents of two patients enrolled who died, presented a claim against the hospital and the study was halted.
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Collaborators: SPANISH HEALTH RESEARCH FUND (FIS) (Unknown)
Responsible Party: Principal Investigator, Antonio Perez-Martinez, Servicio de Hemato-Oncología Pediátrica, Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNJ-NK-01/2009
Record Dates: First submitted 2011-03-25; First posted 2011-04-19 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Childhood Solid Tumor
Keywords: HAPLOIDENTICAL STEM CELL TRANSPLANTATION; NK CELL; IL-15
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IL-15 STIMULATED NK CELLS (Experimental)
  Interventions: Other: HAPLOIDENTICAL IL-15 STIMULATED NK CELLS

INTERVENTIONS:
Other: HAPLOIDENTICAL IL-15 STIMULATED NK CELLS — ONE MEGADOSE 30 DAYS AFTER TRANSPLANTATION (DOSE WILL DEPEND ON PATIENT BODY WEIGHT)
  Other Names: CELL THERAPY

SUMMARY:
The investigators propose a new antitumor cell therapy for treating childhood refractory solid tumours. The aim of this study is explore the graft versus tumour effect mediated by allogenic natural killer cells (NKs). NK cell alloreactivity can be predicted by donor killer immunoglobulin-like receptors (KIRs) and human leukocyte antigen (HLA) class I alleles mismatch. Cells without an inhibitory HLA ligand may trigger natural killer cell activation and elimination of those target cells. Reduced risk of relapsed has been described in malignant cancer after haploidentical stem cell transplantation when HLA ligands against the inhibitory KIRs present in the donor were absent in the recipient (KIR-HLA receptor-ligand mismatch). NK alloreactivity could also be obtained by Natural Killer Receptor (NCR), Toll-Like-Receptors (TLRs) and NKG2D receptor stimulation mediated by cytokines or tumour cell lines.

This will be an open, non randomized, Phase I/II clinical trial, with a double objective: therapeutic exploratory. The investigators aim at studying safety and efficacy of haploidentical stem cell transplantation for the treatment of these malignancies with no cure known. Patients will receive an haploidentical stem cell transplantation, followed by IL-15 stimulated NK cells infusion one month after transplantation. Efficacy of the procedure will be evaluated with up-to-date radiological techniques, molecular studies and functional assays.

DETAILED DESCRIPTION:
The investigators propose a new antitumor cell therapy for treating childhood refractory solid tumours. The aim of this study is explore the graft versus tumour effect mediated by allogenic natural killer cells (NKs). NK cell alloreactivity can be predicted by donor killer immunoglobulin-like receptors (KIRs) and human leukocyte antigen (HLA) class I alleles mismatch. Cells without an inhibitory HLA ligand may trigger natural killer cell activation and elimination of those target cells. Reduced risk of relapsed has been described in malignant cancer after haploidentical stem cell transplantation when HLA ligands against the inhibitory KIRs present in the donor were absent in the recipient (KIR-HLA receptor-ligand mismatch). NK alloreactivity could also be obtained by Natural Killer Receptor (NCR), Toll-Like-Receptors (TLRs) and NKG2D receptor stimulation mediated by cytokines or tumour cell lines.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 22 years.
* Histological solid tumor confirmation.
* Measurable solid tumor by image or molecular techniques.
* Solid tumors that have failed to at least 2 chemotherapy protocols.
* Suitable haploidentical donor available.
* Lansky score > 60%.

Exclusion Criteria:

* Serum bilirubin > 3 mg/dl
* GFR < 40 ml/min/1.73 mw
* Cardiac left ventricular ejection fraction < 40%
* HIV+
* Pregnant
* Unfavorable psycho-social report.
* Antecedent of abandonment treatment.

Ages: 6 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events according to NCI-CTC v3.0 CRITERIA as a measure of safety and tolerability | Up To 1 Year After Transplantation

SECONDARY OUTCOMES:
Objective Response Rate According RECIST V1.1 | Up To One Year After Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO PEREZ-MARTINEZ, MD, PhD, Principal Investigator — HOSPITAL UNIVERSITARIO NINO JESUS
Locations (1):
- Hospital Infantil Universitario Niño Jesus, Madrid, Madrid, Spain

REFERENCES:
- [Background] Perez-Martinez A, Leung W, Munoz E, Iyengar R, Ramirez M, Vicario JL, Lassaletta A, Sevilla J, Gonzalez-Vicent M, Madero L, Diaz-Perez MA. KIR-HLA receptor-ligand mismatch associated with a graft-versus-tumor effect in haploidentical stem cell transplantation for pediatric metastatic solid tumors. Pediatr Blood Cancer. 2009 Jul;53(1):120-4. doi: 10.1002/pbc.21955. PMID 19215002